CLINICAL TRIAL: NCT06288789
Title: Turkish Validity and Reliability of the Social Frailty Index in the Older Adults
Brief Title: Turkish Validity and Reliability of the Social Frailty Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Elif Gur Kabul, Assistant Professor, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SFI-TR
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Elderly; Frailty; Quality of Life
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): 65 years and above older adults
  Interventions: Other: Social Frailty Index

INTERVENTIONS:
Other: Social Frailty Index — Social Frailty Index will be applied twice, one week apart.

SUMMARY:
The aim was to examine the validity and reliability of the Social Frailty Index in Turkish among older adults. 65 years and above older adults will be included included in the study. Older adults who agree to participate in the study will first be administered the Hodkinson Mental Test. Those who score 6 points and above will be included in the study. To evaluate the validity of the "Social Frailty Index", Social Inclusion Scale, Older people's quality of life-brief (OPQOL-brief) and Lubben Social Network Scale will be applied to the participants. To determine the reliability of the "Social Frailty Index", older adults who do not receive any treatment will be tested and re-tested at one-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Getting a score of 6 or above on the Hodkinson Mental Test

Exclusion Criteria:

* -Having another chronic disease that can cause pain
* Having a neurological disease
* Being blind
* Having an orthopedic, neurological or mental disability

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 186 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Social Frailty Index | 10 minutes
  Social Frailty Index included age, gender and eight social predictors

SECONDARY OUTCOMES:
Socıal Inclusıon Scale | 10 minutes
  It consists of 22 items
Older people's quality of life-brief (OPQOL-brief) | 8 minutes
  It consists of 13 items
Lubben Social Network Scale | 5 minutes
  It consists of 6 items

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Gur Kabul, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gur Kabul E, Aksoy CC, Basakci Calik B. The validity of Turkish version of Social Frailty Index in older adults: An index of social attributes predictive of mortality. Rev Esp Geriatr Gerontol. 2025 Mar-Apr;60(2):101556. doi: 10.1016/j.regg.2024.101556. Epub 2024 Oct 19. PMID 39426188